CLINICAL TRIAL: NCT00250406
Title: Assessment of Bacterial Adherence and Biofilm Formation on a Triclosan Loaded Ureteral Stent: A Phase II Study
Brief Title: Assessment of Drug-eluting Ureteral Stent on Bacterial Adherence and Biofilm Formation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, John Denstedt, Chair/Chief, Department of Surgery, Western University, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R-05-646
Record Dates: First submitted 2005-11-04; First posted 2005-11-08 (Estimated); Last update posted 2013-12-20 (Estimated); Status verified 2013-12

CONDITIONS: Renal Calculi; Ureteral Obstruction
Keywords: urolithiasis; ureteral stent; triclosan; drug eluting
MeSH Terms: conditions — Kidney Calculi; Ureteral Obstruction; Urolithiasis | interventions — Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Percuflex Plus Ureteral Stent
  Interventions: Device: Ureteral Stent
- 2 (Experimental): TRIUMPH stent (triclosan-eluting stent)
  Interventions: Device: Ureteral Stent

INTERVENTIONS:
Device: Ureteral Stent — triclosan-eluting ureteral stent
  Other Names: TRIUMPH STENT
  Arms: 2
Device: Ureteral Stent — Percuflex Plus Stent as the control
  Other Names: Percuflex Plus Stent
  Arms: 1

SUMMARY:
The purpose of this study is to determine the clinical effects of a triclosan stent on adherent bacteria, stent biofilms, and patient urine cultures in patients with an indwelling triclosan ureteral stent. The patient populations that will be tested include: patients following ureteroscopy and patients scheduled to undergo shockwave lithotripsy who require a ureteral stent. It is hypothesized that triclosan eluting ureteral stents will reduce the number of bacteria both on (within biofilm) and around (in the urine) a ureteral stent.

ELIGIBILITY:
Inclusion Criteria:

* Patients who undergo ureteroscopy for any reason and require a ureteral stent post-operatively as determined by the surgeon (e.g. renal obstruction, ureteral edema, ureteral perforation, large stone fragments to pass, following ureteral dilation, ureteral trauma, solitary kidney, or any other reason left to the discretion of the surgeon).
* Patients undergoing extracorporeal shockwave lithotripsy (ESWL) who will require a stent as determined by the treating urologist (e.g. solitary kidney, ureteral stone > 1 cm, renal stone > 1.5 cm, significant renal obstruction, history of pyelonephritis, or any other reason left to the discretion of the surgeon).
* Patients who have or are going to have chronic ureteral stents, for any reason.
* Patients willing to return to St. Joseph's Hospital's Urology Clinic for follow-up.

Exclusion Criteria:

* Age ≤ 17 years
* Patients unable to consent.
* Any patient requiring endocarditis or prosthetic device prophylaxis (e.g. fresh arthroplasty etc.).
* Pregnant females
* Immunocompromised patients
* Significant urinary symptoms (urgency, dysuria, strangury, hematuria) or other bladder pathology that may cause these symptoms (e.g. interstitial cystitis)
* Anyone in the investigator's opinion that would be unsuitable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2005-11; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Primary objective is to determine if the number of stent adherent bacteria will be less in patients who receive a triclosan stent compared to a control/standard stent. | at time of intervention

SECONDARY OUTCOMES:
Secondary objectives to be assessed include the amount of biofilm adherent to each stent and each patient's urine culture. | at time of intervention

CONTACTS AND LOCATIONS:
Overall Officials: John D Denstedt, MD, FRCSC, Principal Investigator — St. Joseph's Hospital, The University of Western Ontario
Locations (1):
- Urology, St. Joseph's Hospital, London, Ontario, Canada